CLINICAL TRIAL: NCT04154280
Title: Combination of 68Ga-PSMA PET Data With Magnetic Resonance Spectroscopy Data (MRS) for Evaluating Prostate Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TASMC-19-ES-0590-CTIL
Record Dates: First submitted 2019-10-29; First posted 2019-11-06 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- prostate cancer Patients (Experimental): patients over the age of 18 with diagnosed prostate cancer at different stages of the disease.
  Interventions: Diagnostic Test: PET/MR scan

INTERVENTIONS:
Diagnostic Test: PET/MR scan — * The PET will be performed with 68Ga-PSMA tracer.
  * The 3 tesla magnet of the MRI will be used with sequence allowing MRS acquisition, additional sequences will include T2-weighted contrast and diffusion weighted contrast.
  * Images will be analyzed visually and quantitatively. Quantitative analysis will include MR parameters such as DWI apparent diffusion coefficient (ADC) and PET quantitative metabolic data such as standard uptake values (SUV) or Ki (in case dynamic PET protocol will be applied). In addition, content relationship between metabolic entities detected will be extracted.
  Quantitative data will be correlated to clinical and pathological data to check accuracy, specificity and sensitivity.

SUMMARY:
Prostate cancer is the second most common cancer among man and the fourth most occurring over all . Characterization and management of the diagnosed prostate cancer is a challenging task due to its clinically and morphologically diversity. Clinically, this cancer range from indolent growing slowly malignancy, which does not threatened the patient life, to aggressive tumor that metastasize rapidly with very bad prognosis. Therapy of prostate cancer ranges from a "watch and wait" approach to hormone deprivation therapy to aggressive surgical, radiation, and cryosurgical therapies depending on the cancer characteristics. Prostate cancer is diagnosed using digital rectal examination, serum prostate-specific antigen (PSA) testing and transrectal ultrasonography (US)-guided biopsies . Imaging technologies have been adapted as a non-invasive method to obtain a comprehensive assessment of the disease. MRI is widely used and more specifically multiparameter MRI (mMRI) for detection, staging and tumor localization. mMRI uses multiphase modes including diffusion-weighted and dynamic contrast-enhanced imaging in addition to T2-weighted imaging to identify and classify cancer type . Magnetic Resonance Spectroscopy (MRS) is MRI technique that allow detection of tissue metabolic composition which is occasionally used to characterize prostate cancer, however is not used as a standard procedure. By suppression of water and fat signal, MRS sequence can detect relationship between lower concentration prostatic metabolites such as citrate, choline, creatine, and polyamines in the cell cytosol and in the extra cellular ducts.

Other imaging modalities used to characterize prostate cancer include ultrasound (US), computerized tomography (CT), functional imaging like bone scanning (BS) and hybrid imaging like choline based positron emission tomography and CT (PET/CT). However all of these modalities show disappointing sensitivity .

DETAILED DESCRIPTION:
In recent years a new modality has emerged showing promising accuracy targeting the Prostate Specific Membrane Antigen (PSMA) which is significantly overexpressed in prostate tumor cells. By attaching radioactive isotope 68Ga to PSMA ligands, PET/CT molecular imaging can provide information regarding prostate cancer relapses and metastases with high contrast . Several recent studies showed the potential of 68Ga-PSMA PET in many application correlated with prostate cancer such as staging, identifying reoccurrence, guided biopsy and others . In the study, we wish to utilize the new hybrid PET/MR technology and combine 68Ga-PSMA PET studies with MRS information in order to explore correlation between the data obtained by both modalities and investigate the implication on the disease characteristics.

ELIGIBILITY:
Inclusion Criteria:

1.patients over the age of 18 with diagnosed prostate cancer at different stages of the disease.

Exclusion Criteria:

1. Patients younger than 18 years
2. contraindication to MRI or to intravenous gadolinium injection.

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-04-10 (Estimated); Primary Completion 2021-05-10 (Estimated); Study Completion 2022-04-10 (Estimated)

PRIMARY OUTCOMES:
Patients who preformed 68Ga-PSMA for staging prostate cancer. | 1 year
  Investigate implication of combining 68Ga-PSMA PET data and MRS data on staging and monitoring of prostate cancer

IPD SHARING:
Plan to Share IPD: Undecided